CLINICAL TRIAL: NCT00002347
Title: A Master Protocol to Evaluate the Safety and Efficacy of Multi-Drug Combination Antiretroviral Therapy for the Treatment of HIV Infection: Retrovir/HIVID/Nevirapine and Retrovir/HIVID/Invirase
Brief Title: The Safety and Effectiveness of Retrovir Plus HIVID Combined With Either Nevirapine or Invirase in the Treatment of HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parexel (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 229C; ICC 001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-06

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Nevirapine; Saquinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Saquinavir; Nevirapine; Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Saquinavir
Drug: Nevirapine
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To evaluate the tolerance and immunologic and virologic effects of multidrug combinations of antiretrovirals in patients with HIV infection. Specifically, to evaluate zidovudine/zalcitabine ( AZT / ddC ) alone or in combination with either nevirapine or saquinavir ( Ro 31-8959 ).

Administration of three-drug combinations for treatment of HIV infection is preferred over monotherapy or duotherapy. A system has been designed to rapidly evaluate current multidrug combinations of antiretrovirals and allow the addition of new agents as they become available.

DETAILED DESCRIPTION:
Administration of three-drug combinations for treatment of HIV infection is preferred over monotherapy or duotherapy. A system has been designed to rapidly evaluate current multidrug combinations of antiretrovirals and allow the addition of new agents as they become available.

Patients are randomized to receive AZT/ddC either alone or in combination with nevirapine or Ro 31-8959 for a minimum of 48 weeks. Patients are followed at weeks 2 and 4 and every 4 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Encouraged:

* PCP chemoprophylaxis for patients whose CD4 count falls below 200 cells/mm3 or who develop PCP on study.

Allowed:

* Secondary prophylaxis with nonexperimental agents in patients who develop TB, Mycobacterium avium-intracellulare, toxoplasmosis, histoplasmosis, cryptococcosis, disseminated candidiasis, or cytomegalovirus infection.
* Acyclovir for 21 days or less for acute treatment.
* Recombinant erythropoietin and G-CSF for grade 3 or worse anemia and neutropenia, respectively.

Patients must have:

* HIV infection.
* CD4 count 200 - 500 cells/mm3.
* No prior antiretroviral therapy.
* Life expectancy of at least 48 weeks.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Participating centers are encouraged to enroll female patients.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Any grade 3 or greater toxicity.
* Symptoms of peripheral neuropathy.
* Malabsorption or severe chronic diarrhea.
* Inability to eat at least one meal daily because of chronic nausea, emesis, or abdominal or esophageal discomfort.

Concurrent Medication:

Excluded during the first 28 days of nevirapine administration:

* Augmentin and other antibiotics containing clavulanic acid.

Excluded at any time:

* Dicumarol, warfarin, and other anticoagulant medications.
* Tolbutamide.
* Cimetidine.
* Erythromycin.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* History of grade 2 or worse peripheral neuropathy from any cause.

Prior Medication:

Excluded:

* Any prior antiretroviral therapy.

Excluded within 4 weeks prior to study entry:

* Immunomodulating agents such as systemic corticosteroids, IL-2, alpha-interferon, beta-interferon, or gamma-interferon.
* Immunotherapeutic vaccines.
* Cytotoxic chemotherapy.
* Erythromycin.
* Dicumarol, Coumadin / warfarin, and other anticoagulant medications.
* Phenobarbital.
* Amoxicillin / clavulanate.
* Ticarcillin / clavulanate.
* Tolbutamide.
* Erythromycin.
* Cimetidine.

Prior Treatment:

Excluded within 4 weeks prior to study entry:

* Non-local radiation therapy. Current alcohol or illicit drug use that would interfere with ability to comply with study requirements.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL Intl Corp / InterCo Collaboration Ctr, Waltham, Massachusetts, United States

REFERENCES:
- [Background] Thompson M, Myers M, Salgo M, Rousseau F, Odorisio M, Warburg M. A master protocol to evaluate the safety and efficacy of multidrug combination antiretroviral therapy with zidovudine and zalcitabine with or without saquinavir or nevirapine for the treatment of HIV infection. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:109 (abstract no 242)